CLINICAL TRIAL: NCT00123162
Title: Sildenafil Citrate in the Treatment of Primary Dysmenorrhea
Brief Title: Viagra in the Treatment of Primary Dysmenorrhea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20477
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Dysmenorrhea
Keywords: Sildenafil
MeSH Terms: conditions — Dysmenorrhea | interventions — Sildenafil Citrate; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil Citrate (Experimental): A single vaginal dose of Viagra 100 mg.
  Interventions: Drug: Sildenafil Citrate
- Placebo (Placebo Comparator): A single vaginal dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil Citrate — A single vaginal dose of sildenafil citrate 100 mg and monitored for 4 hours.
  Other Names: Viagra
  Arms: Sildenafil Citrate
Drug: Placebo — A single vaginal dose of placebo and monitored for 4 hours.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The primary hypothesis is that a 100mg single dose of sildenafil citrate (Viagra) will have a higher improvement rate when compared to placebo in the treatment of moderate to severe primary dysmenorrhea.

DETAILED DESCRIPTION:
It is well established that excess prostaglandin production in primary dysmenorrhea leads to ischemia of the uterine muscle, which consequently causes pelvic pain. A large number of drugs have been studied for pain relief in dysmenorrhea patients, with non-steroid anti-inflammatory drugs (NSAIDS) being the most effective with the overall success rate of more than 75%. Sildenafil citrate (Viagra) is an inhibitor that augments the vasodilatory effects of nitric oxide by preventing the degradation of Cyclic guanosine monophosphate (cGMP) in the uterine muscle. Sildenafil is commonly used in the treatment of male erectile dysfunction, pulmonary hypertension in children and adults, and in vitro fertilization. To date it has not been used in the treatment of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Primary dysmenorrhea at current visit, with a visual analogue scale (VAS) score of >35; pain defined as moderate or severe on a categorical of none, mild, moderate, severe.

Exclusion Criteria:

* Secondary dysmenorrhea
* Any current medication
* Serious medical condition

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Legro, M.D., Principal Investigator — Penn State University College of Medicine
Locations (1):
- Nova Gradiska General Hospital, Strossmayerova 17, Zagreb, Croatia

REFERENCES:
- [Derived] Dmitrovic R, Kunselman AR, Legro RS. Sildenafil citrate in the treatment of pain in primary dysmenorrhea: a randomized controlled trial. Hum Reprod. 2013 Nov;28(11):2958-65. doi: 10.1093/humrep/det324. Epub 2013 Aug 6. PMID 23925396

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil Citrate: A single vaginal dose of sildenafil citrate 100 mg.
Period: Overall Study
Arm/Group | Sildenafil Citrate | Placebo
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil Citrate | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (5.7) | 23.3 (4.8) | 23.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Croatia | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Was Total Pain Relief Over 4 Hours (TOPAR4), Comparing a Single Dose of Sildenafil 100 mg to a Single Dose of Placebo.
Description: The Total Pain Relief (TOPAR) Scale rates the level of pain relief on a scale of 0=None, 1=Mild, 2=Moderate, 3=Excellent, 4=Complete. The TOPAR scale was completed each hour after administration of study drug for a total of 4 hours. The 4 hourly scores were summed for a final TOPAR4 score that ranged between 0 and 16, with higher values indicating greater pain relief over time. Missing TOPAR scores after the first hour were imputed using the last-observation-carried-forward approach.
Time Frame: Hours 1, 2, 3 and 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil Citrate | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 11.9 (3.2) | 6.4 (2.1)
Statistical Analysis 1: Comparison: Sildenafil Citrate vs Placebo; With 26 subjects per treatment group and an assumed within-group standard deviation of 7 units, the study was designed to have 90% statistical power for a two-sided, 0.05 significance level test to detect a difference of 6.5 units in TOPAR4 between a single dose of 100 mg of sildenafil and placebo. However, we anticipated subject drop-out as high as 15%; therefore, we planned to recruit 31 subjects per treatment group; Test type: Superiority or Other; p < 0.001, ANCOVA; adjusted for baseline pain intensity (Visual Analog Scale (VAS) score); Mean Difference (Net) = 5.3, 95% CI 2-sided [2.9 to 7.6]

2. Secondary Outcome: Improvement in Pain Severity Determined by Visual Analog Scale (VAS).
Description: The Visual Analog Scale (VAS) assesses pain intensity. The scale is 100 mm long; the extremes of the scale are to the left, "no pain" and to the right, "worst pain I have ever felt." The VAS score is determined by measuring the distance (in mm) from the left side of the scale to the point that the patient marked. The score ranges from 0 to 100, with higher values indicating greater pain.
Time Frame: Each hour of the study (0, 1, 2, 3, 4).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sildenafil Citrate | Placebo
Number analyzed (Participants) | 13 | 12
mm
  Hour 0 | 91.2 (11.2) | 95.6 (5.3)
  Hour 1 | 65.2 (21.2) | 88.6 (10.9)
  Hour 2 | 23.4 (25.3) | 72.5 (11.8)
  Hour 3 | 13.8 (25.3) | 58.5 (19.8)
  Hour 4 | 8.8 (25.0) | 51.4 (26.6)
Statistical Analysis 1: Comparison: Sildenafil Citrate vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Mean Difference (Net) = -42.6, 95% CI 2-sided [-58.3 to -26.8] — Comparison of the VAS score at hour 4 (Sildenafil Citrate - Placebo)

ADVERSE EVENTS:
Arm/Group | Sildenafil Citrate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No